CLINICAL TRIAL: NCT02171819
Title: A Phase 1 Double Blinded, Randomized, Placebo-Controlled Study to Examine the Safety and Immunogenicity of an Inactivated A/H5N1 Influenza Vaccine (IVACFLU-A/H5N1) Produced by IVAC in Healthy Adult Volunteers in Vietnam
Brief Title: Influenza A/H5N1 Vaccine Clinical Trial (IVACFLU-A/H5N1) - Phase 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); World Health Organization (Other); Institut Pasteur (Industry); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: IVAC A/H5N1; VAC021 (Other: PATH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Influenza A Subtype H5N1 Infection
Keywords: Influenza; Avian; H5N1; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IVACFLU-A/H5N1, 7.5 mcg (Experimental): IVACFLU-A/H5N1, 7.5 mcg HA per dose
  Interventions: Biological: IVACFLU-A/H5N1, 7.5 mcg
- IVACFLU-A/H5N1, 15 mcg (Experimental): IVACFLU-A/H5N1, 15 mcg HA per dose.
  Interventions: Biological: IVACFLU-A/H5N1, 15 mcg
- Placebo (Placebo Comparator): Phosphate buffered saline
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: IVACFLU-A/H5N1, 7.5 mcg — Contains 7.5 mcg HA and 0.6 mg of aluminum hydroxide adjuvant per 0.5 mL dose.
  Arms: IVACFLU-A/H5N1, 7.5 mcg
Biological: IVACFLU-A/H5N1, 15 mcg — Contains 15 mcg HA and 0.6 mg of aluminum hydroxide adjuvant per 0.5 mL dose
  Arms: IVACFLU-A/H5N1, 15 mcg
Other: Placebo Comparator — PBS, pH 7.2 in 0.5 mL single-dose vials.
  Other Names: Phosphate Buffered Saline
  Arms: Placebo

SUMMARY:
This is a first-in-human study of safety and immunogenicity of an A/H5N1 inactivated whole cell vaccine when given in two injections in two doses (low and high) compared to a placebo in 76 healthy adult subjects in Vietnam. Vaccine and placebo are manufactured by the IVAC in Vietnam.

DETAILED DESCRIPTION:
This is a phase 1, double blinded, randomized, placebo-controlled study. Seventy-six healthy male and female adults, 18 to 30 years of age, will be enrolled into the trial. Subjects will be randomized to one of three treatment allocations: 32 subjects to 7.5 mcg/dose vaccine (low dose), 32 subjects to 15 mcg/dose vaccine (high dose) and 12 subjects to placebo. This sample size was selected to enable at least 30 evaluable subjects in each of the groups receiving active vaccine. The study will utilize a "block randomization" to assure a balance of 8:8:3 vaccine and placebo when all subjects are enrolled. The study will be double blinded, meaning the study subjects, investigators, and the sponsor will be unaware of the treatment allocated to each subject until the clinical trial database is declared final and locked.

Since this is a first-in-human study, all injections of study product will be sequential and staggered and there will be a safety evaluation between a sentinel cohort of 19 subjects and the remaining 57 study subjects for both the 1st and 2nd doses in the study.

A sentinel group of 19 participants' enrollment and vaccination will precede the remainder of the study group by approximately 2-3 weeks.

Product administration for both injections of vaccine or placebo will be sequential and staggered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 through 30 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* Healthy adults, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits.
* For females, willing to utilize reliable birth control measures (intrauterine device, hormonal contraception, condoms) through the Day 42 visit

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 42 visit.
* Current or recent (within two weeks of enrollment) acute illness with or without fever.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products prior to the Day 42 visit.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, ≥ 0.5 mg per kg per day; topical steroids are allowed.)
* History of asthma.
* Hypersensitivity after previous administration of any vaccine.
* Other AE following immunization, at least possibly related to previous receipt of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Known hypersensitivities (allergies) to food or the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatobiliary, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of any blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressed or immunodeficient condition of any kind.
* Known chronic HBV or HCV infection.
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause.
* History of chronic alcohol abuse and/or illegal drug use.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study product for all women of childbearing potential.)
* History of Guillain-Barré Syndrome
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Le Hoang San, MD, Principal Investigator — Pasteur Institute, Ho Chi Minh City
Locations (1):
- Ben Luc Health Center, Bến Lức, Long An Province, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phan TL, Ho VT, Vu MH, Nguyen TN, Duong HT, Holt R, Wahid R, Donnelly J, Flores J. Clinical testing of an inactivated influenza A/H5N1 vaccine candidate in a double-blinded, placebo-controlled, randomized trial in healthy adults in Vietnam. Vaccine. 2016 Oct 26;34(45):5449-5456. doi: 10.1016/j.vaccine.2016.08.055. Epub 2016 Aug 31. PMID 27591953
- See also: Journal "Vaccine" on line by Elsevier — http://doi.org/10.1016/j.vaccine.2017.03.094
- See also: Results of clinical trial published on line in the journal Vaccine — http://doi.org/10.1016/j.vaccine.2016.08.055

RESULTS

PARTICIPANT FLOW:
Groups:
- IVACFLU-A/H5N1, 7.5 mcg: IVACFLU-A/H5N1, 7.5 mcg HA per dose, given by intramuscular (IM) injection at Day 0 and Day 21.
- IVACFLU-A/H5N1, 15 mcg: IVACFLU-A/H5N1, 15 mcg HA per dose, given IM at Day 0 and Day 21.
- Placebo: phosphate buffered saline, given IM at Day 0 and Day 21.
Period: Overall Study
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Placebo
Started | 31 | 32 | 12
Completed | 31 | 32 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 12 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 12 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 23.7 [19 to 30] | 23.5 [19 to 30] | 23.7 [18 to 28] | 23.6 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 7 | 31
  Male | 20 | 19 | 5 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Kinh | 31 | 32 | 12 | 75
  Khmer | 0 | 0 | 0 | 0
  Hoa | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 31 | 32 | 12 | 75
  Other | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 31 | 32 | 12 | 75

OUTCOME MEASURES:

1. Primary Outcome: Immediate Reactions Occurring Within 60 Minutes of Administration of Any Dose
Description: Data presented are after 1st and 2nd vaccination combined. All participants were observed for immediate reactions for 60 minutes after administration of study product, with appropriate medical treatment readily available in case of an anaphylactic reaction following the administration of study product.
Time Frame: 60 min post injection
Population: Intent to treat population.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Vaccine: Results of low and high doses combined
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With at Least One Solicted Reactogenicity After Both Injections
Description: Data presented are after 1st and 2nd vaccination combined. Solicted reactogenicity are local and systemic events that are expected after injection and specifically asked of the participant. Only reported reactogenicity is presented. If not shown, then no participant reported that reaction in any study group.
  Local reactions are redness, swelling, pain, tenderness, and hardness. Systemic reactions are actual and subjective fever, chills, cough, difficulty breathing, runny nose, nasal congestion, sore throat, hoarseness of voice, headache, confusion. convulsions/seizures, fatigue/malaise, muscle aches (generalized), joint pain, pink or red eyes, sore eyes, itchy eyes, drainage from eyes. ear pain or discharge, rash, abdominal pain, diarrhea, vomiting, and jaundice.
Time Frame: Within 7 days after injection
Population: Participants who were randomized and received study injections
Measure: Count of Participants; unit: Participants
Groups:
- Combined Vaccine: The high- and low-dose vaccine participants combined
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Participants
  Subjects with at least one solicted AE | 26 | 26 | 52 | 4
  Subjects with at least one local solicted AE | 25 | 24 | 49 | 3
  Subjects with at least one systemic solicited AE | 13 | 14 | 27 | 4
  Local reactions--Pain | 18 | 16 | 34 | 1
  Local reactions--Tenderness | 21 | 23 | 44 | 3
  Systemic reactogenicity--Abdominal pain | 1 | 0 | 1 | 0
  Systemic reactogenicity--Chills | 1 | 3 | 4 | 0
  Systemic reactogenicity--Cough | 3 | 2 | 5 | 2
  Systemic reactogenicity--Diarrhea | 0 | 1 | 1 | 0
  Systemic reactogenicity--Ear pain/discharge | 0 | 1 | 1 | 0
  Systemic reactogenicity--Fatigue/Malaise | 3 | 5 | 8 | 2
  Systemic reactogenicity--Fever | 0 | 3 | 3 | 0
  Systemic reactogenicity--Sore eyes | 1 | 0 | 1 | 0
  Systemic reactogenicity--Sore throat | 2 | 2 | 4 | 2

3. Primary Outcome: Number of Participants With at Least One Unsolicited AE
Description: Summary of number of participants with at least one unsolicited AE after 1st and 2nd vaccination combined. Please see the adverse event section of this report for full details.
Time Frame: Within 7 weeks of injection
Population: Intent to treat population. Please see more detail in the AE section of this posting.
  Table 14.2.1.2.1 Summary of Unsolicited Adverse Events by System Organ Class and Preferred Term (After 1st and 2nd Vaccination Combined) Intention-to-Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: phosphate buffered saline, given at Day 0 and Day 21
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Placebo
Number analyzed (Participants) | 31 | 32 | 12
Participants | 12 | 12 | 4

4. Primary Outcome: All Serious Adverse Events (SAEs) Occurring Within 3 Weeks of Receipt of Any Dose
Description: Summary data. Data presented are after 1st and 2nd injections combined. Please see AE reporting section of this report for full details.
Time Frame: Within 3 weeks of any injection
Population: Table 14.2.2.3.1 Summary of Serious Unsolicited Adverse Events by System Organ Class and Preferred Term (After 1st and 2nd Vaccination Combined) Intention-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Placebo
Number analyzed (Participants) | 31 | 32 | 12
Participants | 0 | 0 | 0

5. Secondary Outcome: The Proportion of Subjects Achieving a Hemagglutination Inhibition (HAI) Titer ≥ 1:40 Pre-vaccination (Day 0) to Post 2nd Vaccination (Day 49)
Time Frame: Day 0 to Day 49
Population: Per-protocol analysis set--The Per-Protocol Analysis Set (PPAS) contained all study subjects who received 2 doses of vaccine or placebo and completed the Day 42 visit without major protocol violations that were determined to potentially interfere with immune response to the study vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Vaccine: Low and high dose groups combined
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Participants
  Post vaccination #1 | 7 | 9 | 16 | 0
  Post vaccination #2 | 13 | 18 | 31 | 0

6. Secondary Outcome: The Proportion of Subjects Achieving a Four-fold Rise in HAI Between Doses or From Baseline to Post-Injection 2
Time Frame: Days 21 and 42
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Participants
  Baseline to post 1st vaccination | 11 | 12 | 23 | 0
  From post 1st- to post 2nd vaccination | 9 | 11 | 20 | 0
  Baseline to 2nd vaccination | 21 | 23 | 44 | 0

7. Secondary Outcome: Geometric Mean Titer (GMT) of Hemagglutination Inhibition After Each Dose
Time Frame: Days 0, 21 and 42
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Titers
  Day 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Post vaccination #1 | 12.8 [7.95 to 20.58] | 11.9 [8.17 to 17.31] | 12.3 [9.19 to 16.53] | 5.00 [5.00 to 5.00]
  Post vaccination #2 | 24.5 [15.51 to 38.58] | 27.1 [19.98 to 36.71] | 25.8 [19.77 to 33.57] | 5.00 [5.00 to 5.00]

8. Secondary Outcome: Geometric Mean Titer (GMT) of Neutralizing Antibody After Each Dose
Time Frame: Days 0, 21, and 42
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Combined Vaccine | Placebo
Number analyzed (Participants) | 31 | 32 | 63 | 12
Titers
  Day 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Post vaccination #1 | 9.4 [5.99 to 14.60] | 9.4 [6.52 to 13.46] | 9.4 [7.09 to 12.36] | 5.00 [5.00 to 5.00]
  Post vaccination #2 | 21.9 [13.91 to 34.38] | 23.3 [16.54 to 32.76] | 22.6 [17.16 to 29.70] | 5.00 [5.00 to 5.00]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | IVACFLU-A/H5N1, 7.5 mcg | IVACFLU-A/H5N1, 15 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/12
Other Adverse Events (participants affected / at risk) | 12/31 | 12/32 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVACFLU-A/H5N1, 7.5 mcg (N=31) | IVACFLU-A/H5N1, 15 mcg (N=32) | Placebo (N=12)
Immune system disorders (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Food allergy
Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Urinary tract infection
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Pruritis (itchy skin)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oropharanyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1)
Pyrexia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Apthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No